CLINICAL TRIAL: NCT05622695
Title: Study to Determine if Novel Wearable Monitoring System and Machine-Learning Algorithm Can Model Continuous Pulmonary Artery Pressure Recordings in Human Subjects
Brief Title: Non-invasive Pulmonary Artery Prediction
Acronym: ADOPTS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Silverleaf Medical Sciences INC (Industry)
Collaborators: PIH Health Good Samaritan Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: ADOPTS_GOODSAM
Record Dates: First submitted 2022-11-03; First posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Heart Failure; Pulmonary Arterial Hypertension
MeSH Terms: conditions — Heart Failure; Pulmonary Arterial Hypertension | interventions — Catheterization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Catheterization Arm: Participants will be limited to adults older than 18 years of age, able to consent, planned for the cardiac catheterization lab for a right heart catheterization or in the cardiac care unit with an existing arterial line or Swan-Ganz catheter actively measuring the pulmonary artery pressure on a continuous basis.
  Interventions: Device: catheterization

INTERVENTIONS:
Device: catheterization — Swan-Ganz catheterization (also called right heart catheterization or pulmonary artery catheterization) is the passing of a thin tube (catheter) into the right side of the heart and the arteries leading to the lungs. It is done to monitor the heart's function and blood flow and pressures in and around the heart.

SUMMARY:
Cardiac remote monitoring devices have expanded our ability to track physiological changes used in the diagnosis and management of patients with cardiac disease. Implantable remote monitoring technologies have been shown to predict heart failure events, and guide therapy to reduce heart failure hospitalizations. The CardioMEMs System, the most studied and established remote monitoring system, relies on a pulmonary artery implant for continuous PAP measurement. However, there are no commercially available wearable systems that can reproduce continuous PAP tracings.

This study aims to determine if a machine-learning algorithm with data from a wearable cardiac remote-monitoring system incorporating EKG, heart sounds, and thoracic impedance can reproduce a continuous PAP tracing obtained during right heart catheterization.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age 18+ years
2. Undergoing a right heart cardiac catheterization or in the cardiac care unit with active monitoring using an arterial line or Swan-Ganz catheter.

Exclusion Criteria:

1. Vulnerable population
2. Unable to consent for any reason
3. Unstable patient
4. Known skin reaction to latex or adhesives

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with heart failure conditions.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-10-30 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
The correlation of pulmonary artery pressure values measured by Sawn Gan catheter and that derived by a machine learning algorithm | the Swan-Ganz catheter obtains the pulmonary artery pressures for a minimum of 5 minutes.
  The primary objective of this study is to determine if a machine-learning algorithm with data from a wearable device can reproduce simultaneous pulmonary artery pressure obtained during right heart catheterization or data obtained from a Sawn Ganz catheter already in place in the setting of cardiac care unit admission.
The correlation of pulmonary artery wedge pressure values measured by Sawn Gan catheter and that derived by a machine learning algorithm | the Swan-Ganz catheter obtains wedge pressures first for a minimum of 20 seconds (20-30 seconds).
  The second objective of this study is to determine if a machine-learning algorithm with data from a wearable device can reproduce simultaneous pulmonary artery wedge pressure obtained during right heart catheterization or data obtained from a Sawn Ganz catheter already in place in the setting of cardiac care unit admission.

CONTACTS AND LOCATIONS:
Overall Officials: Jianwei Zheng, Ph.D., Study Chair — Silverleaf Medical Sciences; Ihab Alomari, Dr., Principal Investigator — PIH Good Samaritan Hospital; Islam Abudayyeh, Dr., Study Director — Loma Linda University Health
Locations (1):
- PIH Good Samaritan Hospital, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zheng J, Abudayyeh I, Mladenov G, Struppa D, Fu G, Chu H, Rakovski C. An artificial intelligence-based noninvasive solution to estimate pulmonary artery pressure. Front Cardiovasc Med. 2022 Aug 24;9:855356. doi: 10.3389/fcvm.2022.855356. eCollection 2022. PMID 36093166